CLINICAL TRIAL: NCT05328375
Title: Implementing Telehealth-enhanced Hybrid Cardiac Rehabilitation (THCR) Among Acute Coronary Syndrome Survivors: A Pilot Randomized Controlled Trial
Brief Title: Telehealth-enhanced Hybrid Cardiac Rehabilitation Among Acute Coronary Syndrome Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Andrea Duran, Assistant Professor in the Department of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAT7922 - pilot; KL2TR001874 (NIH)
Record Dates: First submitted 2022-04-01; First posted 2022-04-14 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction
Keywords: Acute Coronary Syndrome; Myocardial Infarction; Cardiac Rehabilitation; Feasibility; Adherence
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth-enhanced Hybrid CR (Experimental): Participants will receive a hybrid version of cardiac rehabilitation.
  Interventions: Behavioral: Telehealth-enhanced Hybrid CR
- Traditional CR (Active Comparator): Participants will receive a standard of care version of cardiac rehabilitation.
  Interventions: Behavioral: Traditional CR

INTERVENTIONS:
Behavioral: Telehealth-enhanced Hybrid CR — Participants in this group attend a total of 24 CR sessions (5 clinic-based + 19 home-based) over a 12-week period. Clinic-based sessions occur during the first week of the program and at the end of each month. Home-based sessions take place remotely once or twice per week via telehealth, depending on the week of the program. Patients are provided with onboarding sessions, remote patient monitoring devices (tablet, pulse oximeter, blood pressure monitor and cuff) and home-based exercise equipment (e.g., stationary bike and weights). Each CR session (clinic and home) is 60 minutes in duration and includes aerobic and resistance exercise training. Patients will also be asked to complete educational videos, as well as document their physical activity, dietary intake, medication management and homework sessions via surveys. Patients will be encouraged (but not required) to achieve ≥30 minutes of moderate aerobic activity, such as brisk walking, on ≥5 days per week.
  Arms: Telehealth-enhanced Hybrid CR
Behavioral: Traditional CR — Participants in this group attend a total of 24 clinic-based CR sessions according to standard of care protocols over a 12-week period. Each CR session is 60 minutes in duration and includes aerobic and resistance exercise training. In addition to scheduled sessions, patients will be asked to complete educational videos, as well as document their physical activity, dietary intake, medication management and homework sessions via surveys. Patients will be encouraged (but not required) to achieve ≥30 minutes of moderate aerobic activity, such as brisk walking, on ≥5 days per week.
  Arms: Traditional CR

SUMMARY:
This study investigates the feasibility of conducting a randomized controlled trial of telehealth-enhanced hybrid cardiac rehabilitation (THCR) compared with traditional cardiac rehabilitation (CR) among acute coronary syndrome (ACS) survivors. THCR is a novel, hybrid model that targets the same core components as traditional CR (e.g., exercise training, patient education, and risk factor management), but uses a mixture of telehealth, clinic-, and home-based activities to offer 24 CR sessions (5 clinic-based + 19 home-based) over 12 weeks.

Pilot study ran from March 2022 to May 2023. In 2023, intervention became unavailable, due to a telehealth vendor transition across the implementation site's healthcare system, which necessitated new remote patient monitoring platform to offer the experimental arm. Therefore, the study completed with 10 accrued.

DETAILED DESCRIPTION:
Cardiac Rehabilitation (CR) is a Class I, Level A secondary prevention program that significantly reduces reinfarction and mortality rates in acute coronary syndrome (ACS) survivors. Yet, fewer than 30% of eligible cardiac patients participate in and adhere to CR programs in the United States. One promising avenue for increasing CR participation and adherence is a telehealth-enhanced hybrid CR (THCR) model that combines telehealth, clinic- and home-based CR. Several expert groups have strongly endorsed hybrid CR models that integrate telehealth (i.e., mobile apps, remote monitoring devices) because of their ability to offer the "best of both worlds" (i.e., in-clinic supervision/safety and at-home convenience) while also promoting real-time patient-provider communication and reimbursement as a telemedicine service. Despite its potential, the feasibility of and degree to which THCR improves adherence (e.g., # of completed sessions) and clinical outcomes (e.g., functional capacity) relative to traditional CR requires additional investigation. To understand the feasibility of THCR, the investigator will conduct a single center, two-arm, 1:1 parallel group randomized pilot study comparing THCR with traditional CR among ACS patients (N=40) to evaluate the feasibility (e.g., recruitment, adherence) of conducting an adequately powered randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. over the age of 18;
2. can speak and read English or Spanish;
3. confirmed ACS based on ICD-10 codes; and
4. had their index event within the past 12 months.

Exclusion Criteria:

1. severe disabling chronic medical and/or psychiatric comorbidities determined on a case-by-case basis that prevent safe or adequate participation;
2. high-risk for adverse exercise-related cardiovascular events according to the AACVPR risk stratification criteria;
3. participated in >1 CR program session;
4. deemed unable to comply with the protocol (either self-selected or indicated during screening that s/he could not complete all requested tasks). This includes, but is not limited to, patients with a level of cognitive impairment indicative of dementia, patients with current alcohol or substance abuse, patients with a significant movement or balance disorder that interferes with walking, patients with impaired circulation or poor perfusion that may impede pulse oximeter readings, and patients with severe mental illness (e.g., schizophrenia);
5. home-based environment deemed incompatible with the protocol and/or that prevent safe or adequate participation (either self-selected or indicated during screening/onboarding process); and
6. unavailable for follow-up for reasons such as terminal illness and imminent plans to leave the United States (as we have migrant or mobile patients due to their citizenship and work issues).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea T Duran, PhD, Principal Investigator — Columbia University; Daichi Shimbo, MD, Study Director — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ritchey MD, Maresh S, McNeely J, Shaffer T, Jackson SL, Keteyian SJ, Brawner CA, Whooley MA, Chang T, Stolp H, Schieb L, Wright J. Tracking Cardiac Rehabilitation Participation and Completion Among Medicare Beneficiaries to Inform the Efforts of a National Initiative. Circ Cardiovasc Qual Outcomes. 2020 Jan;13(1):e005902. doi: 10.1161/CIRCOUTCOMES.119.005902. Epub 2020 Jan 14. PMID 31931615
- [Background] Thomas RJ, Beatty AL, Beckie TM, Brewer LC, Brown TM, Forman DE, Franklin BA, Keteyian SJ, Kitzman DW, Regensteiner JG, Sanderson BK, Whooley MA. Home-Based Cardiac Rehabilitation: A Scientific Statement From the American Association of Cardiovascular and Pulmonary Rehabilitation, the American Heart Association, and the American College of Cardiology. Circulation. 2019 Jul 2;140(1):e69-e89. doi: 10.1161/CIR.0000000000000663. Epub 2019 May 13. PMID 31082266
- [Background] Amsterdam EA, Wenger NK, Brindis RG, Casey DE Jr, Ganiats TG, Holmes DR Jr, Jaffe AS, Jneid H, Kelly RF, Kontos MC, Levine GN, Liebson PR, Mukherjee D, Peterson ED, Sabatine MS, Smalling RW, Zieman SJ; ACC/AHA Task Force Members. 2014 AHA/ACC guideline for the management of patients with non-ST-elevation acute coronary syndromes: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Dec 23;130(25):e344-426. doi: 10.1161/CIR.0000000000000134. Epub 2014 Sep 23. No abstract available. PMID 25249585
- [Background] Smith SC Jr, Benjamin EJ, Bonow RO, Braun LT, Creager MA, Franklin BA, Gibbons RJ, Grundy SM, Hiratzka LF, Jones DW, Lloyd-Jones DM, Minissian M, Mosca L, Peterson ED, Sacco RL, Spertus J, Stein JH, Taubert KA; World Heart Federation and the Preventive Cardiovascular Nurses Association. AHA/ACCF Secondary Prevention and Risk Reduction Therapy for Patients with Coronary and other Atherosclerotic Vascular Disease: 2011 update: a guideline from the American Heart Association and American College of Cardiology Foundation. Circulation. 2011 Nov 29;124(22):2458-73. doi: 10.1161/CIR.0b013e318235eb4d. Epub 2011 Nov 3. No abstract available. PMID 22052934
- [Background] Imran HM, Baig M, Erqou S, Taveira TH, Shah NR, Morrison A, Choudhary G, Wu WC. Home-Based Cardiac Rehabilitation Alone and Hybrid With Center-Based Cardiac Rehabilitation in Heart Failure: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2019 Aug 20;8(16):e012779. doi: 10.1161/JAHA.119.012779. Epub 2019 Aug 17. PMID 31423874

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telehealth-enhanced Hybrid CR | Traditional CR
Started | 5 | 5
Completed | 5 | 4 (Participant moved out of state. Prior to formally withdrawing from the study, the participant completed the post-intervention assessments that could be conducted remotely (e.g., feasibility of intervention measure) but did not complete assessments administered as standard of care in the clinic (e.g., 6MWT, DUKE questionnaire).)
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telehealth-enhanced Hybrid CR | Traditional CR | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.1 (10.8) | 63.2 (12.6) | 61.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 3 | 1 | 4
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: Participants]
  United States | 5 | 5 | 10
Six Minute Walk Test Distance [Mean (Standard Deviation); unit: meters] | 501.7 (113.7) | 452.4 (133.7) | 477.0 (119.8)
Health-related Quality of Life Score [Mean (Standard Deviation); unit: score on a scale] | 78.0 (11.2) | 81.3 (12.6) | 79.7 (11.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Successfully Enrolled Into the Pilot Study Per Month
Description: As a measure of enrollment feasibility, the investigator will assess the number of participants who completed recruitment activities and were successfully consented and enrolled into the pilot study per month.
Time Frame: During enrollment, 11 months
Measure: Mean (Standard Error); unit: Participants enrolled per month
Groups:
- All Pilot Study Enrollments: All participants who successfully enrolled into the pilot study
Arm/Group | All Pilot Study Enrollments
Number analyzed (Participants) | 10
Participants enrolled per month | 0.91 (0.21)
Statistical Analysis 1: Comparison: All Pilot Study Enrollments; Test type: Other; Mean = 0.91, 95% CI 1-sided [lower limit 0.62] — The estimate is based on the number of participants enrolled per month over the 11-month recruitment period of the trial. A 1-sided 95% lower confidence limit was computed

2. Primary Outcome: Mean Proportion of CR Sessions Completed by Participants Allocated to the THCR Intervention
Description: As a measure of THCR adherence, the investigator will assess the proportion of CR sessions completed by participants allocated to the THCR intervention, which includes 19 home-based + 5 clinic-based sessions.
Time Frame: Assessed after enrollment (baseline) and until pilot study completion (approximately 12 weeks)
Measure: Mean (Standard Error); unit: Proportion of CR Sessions Completed
Arm/Group | Telehealth-enhanced Hybrid CR
Number analyzed (Participants) | 5
Proportion of CR Sessions Completed | 0.87 (0.13)
Statistical Analysis 1: Comparison: Telehealth-enhanced Hybrid CR; Test type: Other; Mean = 0.87, 95% CI 1-sided [lower limit 0.66] — The estimate is based on the mean proportion of cardiac rehabilitation sessions completed by THCR participants. A 1-sided 95% lower confidence limit was computed

3. Secondary Outcome: Proportion of Participants That Attend ≥1 CR Session After Randomization in Each Arm
Description: This is to assess the feasibility of program initiation among participants allocated to each arm. Participants who attended more than 1 CR session will be tallied. Numerator = total number of participants randomized into each arm who attended at least 1 CR session. Denominator = total number of participants randomized into each arm.
Time Frame: During 12-week follow-up period (Up to 12 weeks)
Measure: Number; unit: proportion of participants
Arm/Group | Telehealth-enhanced Hybrid CR | Traditional CR
Number analyzed (Participants) | 5 | 5
proportion of participants | 1.00 | 1.00
Statistical Analysis 1: Comparison: Telehealth-enhanced Hybrid CR; Test type: Other; Proportion = 1.0, 95% CI 1-sided [lower limit 0.55] — The estimate is based on the proportion of participants in the Telehealth-enhanced Hybrid CR arm who attended at least one cardiac rehabilitation session after randomization. A 1-sided 95% lower confidence limit was computed
Statistical Analysis 2: Comparison: Traditional CR; Test type: Other; Proportion = 1.0, 95% CI 1-sided [lower limit 0.55] — The estimate is based on the proportion of participants in the Traditional CR arm who attended at least one cardiac rehabilitation session after randomization. A 1-sided 95% lower confidence limit was computed

4. Secondary Outcome: Mean Proportion of CR Sessions Completed by Those Allocated to the Traditional CR Intervention
Description: As a measure of traditional CR adherence, the investigator will assess the proportion of CR sessions completed by those allocated to the traditional CR intervention, which includes 24 clinic-based sessions.
Time Frame: Assessed after enrollment (baseline) and until pilot study completion (approximately 12 weeks)
Measure: Mean (Standard Error); unit: Proportion of CR Sessions Completed
Arm/Group | Traditional CR
Number analyzed (Participants) | 5
Proportion of CR Sessions Completed | 0.69 (0.19)
Statistical Analysis 1: Comparison: Traditional CR; Test type: Other; Mean = 0.69, 95% CI 1-sided [lower limit 0.40] — The estimate is based on the mean proportion of cardiac rehabilitation sessions completed by participants in the Traditional CR arm. A 1-sided 95% lower confidence limit was computed

5. Secondary Outcome: Proportion of Participants Who Report Adequate Feasibility of the THCR Intervention
Description: This outcome assesses the proportion of participants in the THCR arm who report an average score ≥4 on the Feasibility of Intervention Measure (FIM), a 4-item scale evaluating patient-perceived feasibility of the intervention. Each item is rated on a 5-point Likert scale ranging from 1 ("strongly disagree") to 5 ("strongly agree"). Individual item scores are summed (possible range: 4 to 20) and averaged (possible range: 1 to 5). Participants with a mean score ≥4 ("agree" or "strongly agree" on average) are considered to perceive the intervention as adequately feasible. Higher scores indicate greater feasibility.
Time Frame: At study completion (approximately 12 weeks)
Measure: Number; unit: Proportion of participants
Arm/Group | Telehealth-enhanced Hybrid CR
Number analyzed (Participants) | 5
Proportion of participants | 1.00
Statistical Analysis 1: Comparison: Telehealth-enhanced Hybrid CR; Test type: Other; Proportion = 1.00, 95% CI 1-sided [lower limit 0.55] — Adequate feasibility was defined as a mean score ≥4 across four post-program items. A 1-sided 95% lower confidence limit was calculated

6. Other Pre Specified Outcome: Change in Total Distance Traveled in 6MWT
Description: This is to measure pre-to-post program change in functional capacity (using the six-minute walk test [6MWT]) among THCR and, separately, traditional CR participants. The 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. The total distance (meters) traveled over a time period of six minutes is used as the outcome by which to compare changes in performance capacity.
Time Frame: Baseline and 3-month post program completion (Week 12)
Population: Excludes one Traditional CR participant who moved out of state and did not complete the post-program 6MWT.
Measure: Mean (Standard Error); unit: distance traveled (meters)
Arm/Group | Telehealth-enhanced Hybrid CR | Traditional CR
Number analyzed (Participants) | 5 | 4
distance traveled (meters) | 27.12 (8.13) | 71.10 (10.30)

7. Other Pre Specified Outcome: Change in Health-related Quality of Life Score
Description: This is to measure pre-to-post program change in health-related quality of life (Duke health profile questionnaire [DUKE; physical, mental, social, and general health composite scores]) among THCR and, separately, traditional CR participants (composite score). The DUKE is a 17-item self-report questionnaire for measuring generic health-related quality of life over a 1-week time period. Responses are scored to calculate physical health, mental health, and social health scores, which are then summed and divided by 3 to obtain a general health score. The general health score ranges from 0 - 100, with high scores indicating better health-related quality of life.
Time Frame: Baseline and 3-month post program completion (Week 12)
Population: Excludes two Traditional CR participants: one who moved out of state and did not complete the post-program in-clinic assessments, and one who did not complete the post-program HRQOL assessment.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Telehealth-enhanced Hybrid CR | Traditional CR
Number analyzed (Participants) | 5 | 3
score on a scale | 1.3 (3.4) | 7.8 (1.1)

ADVERSE EVENTS:
Time Frame: Throughout study duration, approx 14 months
Arm/Group | Telehealth-enhanced Hybrid CR | Traditional CR
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telehealth-enhanced Hybrid CR (N=5) | Traditional CR (N=5)
Low hemoglobin level (Investigations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
In 2023, the study was paused due to a system-wide telehealth vendor transition that disrupted access to the remote patient monitoring platform supporting the Telehealth-Enhanced Hybrid Cardiac Rehabilitation intervention. This disruption limited our ability to enroll participants over the intended 2-year period, and the study ultimately closed with 10 participants enrolled over an 11-month period of active enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT05328375/Prot_SAP_000.pdf